CLINICAL TRIAL: NCT01164852
Title: Expectant Management of Severe Preeclampsia at 28 to 33 Week's Gestation:a Randomized Controlled Trial
Brief Title: Aggressive Versus Expectant Management of Severe Preeclampsia Remote From Term
Acronym: MEXPRE-Latin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complejo Hospitalario Dr. Arnulfo Arias Madrid (Other)
Responsible Party: Principal Investigator, Paulino Vigil-De Gracia, Paulino Emilio Vigil De Gracia, Complejo Hospitalario Dr. Arnulfo Arias Madrid
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ComplejoH 01
Record Dates: First submitted 2010-07-15; First posted 2010-07-19 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Parturition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expectant management (No Intervention): Expectant management: refers to pregnancy prolongation during which time women and fetuses are carefully monitored for indications for delivery.
- Interventionist management (Active Comparator): Interventionist management: in which blood pressure is stabilized, corticosteroids are given for acceleration of fetal maturity and delivery is planned within 48-72 hours.
  Interventions: Procedure: Delivery

INTERVENTIONS:
Procedure: Delivery — Termination of pregnancy (delivery)after completed corticosteroids
  Other Names: Severe preeclampsia; expectant management of severe preeclampsia
  Arms: Interventionist management

SUMMARY:
How best to manage preeclampsia remote from term is controversial because of conflicting maternal and neonatal risks. Gestational age is the most important determinant of neonatal outcome. There are two basic approaches when delivery is not clear indicated by assessment of maternal and fetal well-being. The interventionist care when the delivery is planned within 48 hours and the expectant care which refers to pregnancy prolongation during which time women and fetuses are carefully monitored for indications for delivery.

The purpose of this study is to evaluate maternal and perinatal outcomes with expectant vs interventionist or aggressive management of severe preeclampsia at 28 to 33 weeks of gestation.

DETAILED DESCRIPTION:
Severa Preeclampsia between 28 and 33 weeks of gestation Women and fetus with stable condition All women receive complete dosis of steroids

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy with severe preeclampsia and 28 to 33 weeks of gestation

Exclusion Criteria:

* Uncontrollable blood pressure or persistent severe hypertension (160/110 mmHg)
* Persistent symptoms of preeclampsia
* Maternal complications (HELLP syndrome, acute renal insufficiency, cerebral edema, eclampsia, pulmonary edema)
* Fetal death, restriction of fetal grown

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Perinatal death | After begining the randomization until 4 weeks after delivery.
  Number of perinatal in each group (interventionist or expectant management)

SECONDARY OUTCOMES:
Perinatal complications and maternal complications | Maternal and perinatal complication after begining the randomization until 4 weeks after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Paulino Vigil-De Gracia, MD, Principal Investigator — Complejo Hospitalario; Jack Ludmir, MD, Study Chair — Pennsylvania Hospital
Locations (8):
- Ecuador (2):
  - Hospital Terodoro Maldonado, del IESS, Gauyas
  - Hospital Carlos Andrade Marin, Quito
- Hospital de Gineco-Obstetricia del seguro social, Guatemala City, Guatemala
- Hospital de Ginecologia del Instituto Materno Infantil, Toluca, Mexico
- Panama (2):
  - Complejo Hospitalario Caja de Seguro Social, Panama City, Provincia de Panamá
  - Hospital Santo Tomás, Panama City
- Hospital Nacional Madre Niño, Lima Perú, Lima, Peru
- Hospital Nuestra Señora de Chiquinquira, Maracaibo, Maracaibo, Venezuela